CLINICAL TRIAL: NCT02148484
Title: Comparing Behavioral Therapies for Treating Adolescents With Post-Traumatic Stress Disorder Related to Sexual Abuse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 804439; NCT00417300 (obsolete NCT alias)
Record Dates: First submitted 2013-07-18; First posted 2014-05-28 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: PTSD
Keywords: PTSD; Cognitive Behavioral Treatment; Child Sexual Abuse
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Person-Centered Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Prolonged exposure for adolescents
  Interventions: Behavioral: Prolonged Exposure for Adolescents
- 2 (Active Comparator): Client centered therapy
  Interventions: Behavioral: Client Centered Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure for Adolescents
  Arms: 1
Behavioral: Client Centered Therapy
  Arms: 2

SUMMARY:
Posttraumatic stress disorder (PTSD) is the most common disorder among childhood sexual abuse survivors and is associated with substantial psychosocial and medical problems, but evidence-based treatment for PTSD in adolescents is lacking. This study aims to examine the efficacy and effectiveness of prolonged exposure therapy for adolescents with client-centered therapy.

ELIGIBILITY:
Inclusion Criteria: female gender, age 13-18, and a primary DSM-IV-TR diagnosis of chronic or subthreshold PTSD related to sexual assault

Exclusion Criteria: current suicidal ideation with intent, uncontrolled bipolar disorder, schizophrenia, other thought disorders, or conduct disorder, the presence of a pervasive developmental disorder, initiation of treatment with psychotropic medication within the previous 12 weeks, and current inpatient psychiatric treatment

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2006-02; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline on PTSD symptoms utilizing the Child PTSD Symptom Scale-Interview (CPSS-I) | Baseline, mid-treatment, post-treatment, 3-, 6-, and 12-month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Edna B Foa, Ph.D., Principal Investigator — University of Pennsylvania

REFERENCES:
- [Derived] Chang C, Kaczkurkin AN, McLean CP, Foa EB. Emotion regulation is associated with PTSD and depression among female adolescent survivors of childhood sexual abuse. Psychol Trauma. 2018 May;10(3):319-326. doi: 10.1037/tra0000306. Epub 2017 Jul 6. PMID 28682105
- [Derived] Kaczkurkin AN, Asnaani A, Zhong J, Foa EB. The Moderating Effect of State Anger on Treatment Outcome in Female Adolescents With PTSD. J Trauma Stress. 2016 Aug;29(4):325-31. doi: 10.1002/jts.22116. Epub 2016 Jul 26. PMID 27459380
- [Derived] Foa EB, McLean CP, Capaldi S, Rosenfield D. Prolonged exposure vs supportive counseling for sexual abuse-related PTSD in adolescent girls: a randomized clinical trial. JAMA. 2013 Dec 25;310(24):2650-7. doi: 10.1001/jama.2013.282829. PMID 24368465